CLINICAL TRIAL: NCT05500534
Title: Exploratory Feasibility Study of a Novel Laser System for Endoscopic Disintegration of Urinary Stones With Automatic Real-time Stone Recognition
Brief Title: TELAXMAN - Laser Lithotripsy With Automatic Real-time Stone Recognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LISA Laser Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TELAXMAN
Record Dates: First submitted 2022-08-09; First posted 2022-08-15 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Lithotripsy, Laser
MeSH Terms: interventions — Lithotripsy, Laser

STUDY DESIGN:
Intervention Model Description: Study participants will be scheduled for laser lithotripsy using the investigational device. A comparator arm will also be included, being composed of retrospective, anonymised and non-study related data of patients who underwent laser lithotripsy with a device used in routine lithotripsy interventions at the investigational site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RevoLix HTL+ (Experimental): Laser lithotripsy using the RevoLix HTL+ with active stone recognition
  Interventions: Device: Laser lithotripsy with stone recognition
- Historic control group (Other): Laser lithotripsy without active stone recognition
  Interventions: Other: Laser lithortripsy

INTERVENTIONS:
Device: Laser lithotripsy with stone recognition — Application of Revolix HTL+ which features automatic real-time stone recognition
  Arms: RevoLix HTL+
Other: Laser lithortripsy — Standard laser lithotripsy
  Arms: Historic control group

SUMMARY:
Urolithiasis is an extremely common disease affecting about 12% of the world population with increasing tendency. Urinary stones are sediments that form in the kidney from crystals, such as calcium oxalate.

Currently, urological endoscopy with laser lithotripsy represents the leading and most frequently used method for the treatment of urinary stones of different localization, size and composition.

Surgical urology, including interventional stone treatment, is highly inﬂuenced by technology. With regard to fragmentation properties and effectiveness for all stone types Holmium:yttrium-aluminium-garnet (Ho:YAG) laser lithotripsy has become the standard technology to disintegrate urinary calculi.

In addition, other kinds of lasers are emerging, such as the thulium fiber laser (TFL); a new solid-state, diode-pumped laser that may provide urologists with increased options for stone treatment.

While urolithiasis treatment in general and laser lithotripsy in specific rarely goes along with major complications, recent studies have shown that there are possible indirect risks to the treatment with lasers, such as thermal damages to the urinary tract even at low-power settings if inadequate irrigation is applied. Sufficient irrigation is mandatory to perform safe Ho:YAG laser lithotripsy.

The RevoLix HTL+ automatic real-time stone detection module was developed to overcome these limitations and improve the safety of the patient with regard to potential thermal damages.

The objective of this clinical investigation is to assess the feasibility of stone recognition and disintegration with the RevoLix HTL+ in clinical conditions and to identify hypotheses to be used in future clinical investigations.

ELIGIBILITY:
Inclusion Criteria:

* Subject scheduled for laser lithotripsy
* Subject aged 18 or older
* Subject able to give consent
* Informed consent documented by signature

Exclusion Criteria:

* Subject pregnant or nursing
* Subject requiring emergency lithotripsy
* Contraindication for the surgical procedure:

  * Positive urine culture,
  * Unfit for general anesthesia,
  * Therapeutic anticoagulation, or systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Visual assessment of stone-free status; | During the procedure of laser lithotripsy, which should last for a maximum of 5 hours
  Before retracting the ureteroscope, the surgeon will visualize the postoperative ureter along its entire length and record the stone-free status in the CRF, using the following scale:
  0 - No residue
  1. - Residual fragments ≤4mm
  2. - Residual fragments >4mm Stone-free status is the state-of-the-art methodology for the description of the lithotripsy procedure, which is performed routinely at the investigation site. It does not require any additional invasive testing or procedures and it is performed intra-operatively.
Visual assessment of stone, tissue and endoscope recognition accuracy during laser lithotripsy | During the procedure of laser lithotripsy, which should last for a maximum of 5 hours
  During the procedure, the surgeon will record every incidence of misrecognition by the RevoLix HTL+. Misrecognition is defined as inadequate laser pulse release on healthy tissue or endoscope.
Safety of device - assessment of device deficiencies | During laser lithotripsy (duration of max 5 hours)
  Safety of the device shall be evaluated by systematically reporting DDs and by monitoring the frequency and incidence of these events
Safety of device - assessment of adverse events during the intervention | During laser lithotripsy (duration of max 5 hours)
  Safety of the device shall be evaluated by systematically reporting AEs and SAEs and by monitoring the frequency and incidence of these events
Safety of device - assessment of adverse events during the follow up time | During the follow up time (up to 3 months)
  Safety of the device shall be evaluated by systematically reporting AEs and SAEs and by monitoring the frequency and incidence of these events
New risk identification during the intervention | Within 12 hours after the intervention
  The practitioner will be asked to identify any new risks arising during laser lithotripsy using the investigational device
New risk identification during the follow up time | During the follow up time (up to 3 months)
  The practitioner will be asked to identify any new risks related to the investigational device during the follow up time

SECONDARY OUTCOMES:
Total laser emitted energy (J) | Immediately (up to 1 hour) after the end of the intervention
  Total laser emitted energy is recorded by the laser system during each procedure. This data will be extracted after each procedure for the investigational arm and at the end of the investigation for the matching control arm.
Procedure duration (min) | Immediately (up to 1 hour) after the end of the intervention
  Procedure duration will be recorded in the CRF as the time from endoscope insertion to retraction (Schnitt-Naht Zeit).
PULS classification of potential lesions visible via endoscopy immediately after the procedure | During the procedure of laser lithotripsy, which should last for a maximum of 5 hours
  Before retracting the ureteroscope, the surgeon will visualize the postoperative ureter along its entire length and record PULS classification in the CRF.
  PULS is a 5 grades scale (0 - No lesion; 1 - Superﬁcial mucosal lesion and/or signiﬁcant mucosal oedema/hematoma; 2 - Submucosal lesion; 3 - Perforation with less than 50% partial transection; 4 - Perforation with more than 50% partial transection; 5 - Complete transection), in which lesions are graded independently of their location and extent. In case of multiple lesions, the most severe grading is applied.
Usability and workflow assessment (surgeon's questionnaire) | Within 12 hours after the intervention
  Immediately after his/her first procedure with RevoLix HTL+, the surgeon will fill in a questionnaire regarding the different aspects of the laser system.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schönthaler, Prof. Dr., Principal Investigator — Universitätsklinikum Freiburg
Locations (1):
- Universitätsklinikum Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No